CLINICAL TRIAL: NCT05182892
Title: REducing SPEECH-related Side-effects of Deep Brain Stimulation in Parkinson's Disease Via Automated Speech Analysis
Acronym: RESPEECH-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 2021-01787
Record Dates: First submitted 2021-12-22; First posted 2022-01-10 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Deep brain stimulation; Speech; Dysarthria; Automated speech analysis
MeSH Terms: conditions — Parkinson Disease; Speech; Dysarthria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Speech ratings in part 3 will be performed by speech therapists. They are blinded towards stimulator setting and visit number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: All participants (Experimental): All participants who will participate in part 1.
  Interventions: Other: Change of stimulation amplitudes in dopaminergic OFF drug state
- Part 2: All participants (No Intervention): All participants who participated in part 1
- Part 3: All participants (No Intervention): All participants who will participate in part 3

INTERVENTIONS:
Other: Change of stimulation amplitudes in dopaminergic OFF drug state — Change of stimulation amplitudes during experiment in dopaminergic OFF drug state.
  Arms: Part 1: All participants

SUMMARY:
The investigators' objective is to improve L-dopa sensitive PD-related dysarthria and at the same time reduce DBS-induced speech disorders with the help of automated acoustic analysis in patients with STN-DBS-induced dysarthria.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) of the subthalamic nucleus (STN) is an effective treatment of L-dopa sensitive motor symptoms of Parkinson's disease (PD) but its effects on speech are equivocal. Although some aspects of speech might improve with STN-DBS, stimulation-induced dysarthria represents one of the most common side effects, with a prevalence of up to 90%. Worsening of speech can neutralize the motor benefits of STN-DBS in terms of overall benefit in quality of life. STN-DBS induced dysarthria is not understood in sufficient detail that would allow its prevention or sustained reduction. The human ear is too limited in quantifying subtle changes in speech and to differentiate between parkinsonian and stimulation induced dysarthria. The investigators' objective is to improve L-dopa sensitive PD-related dysarthria and at the same time reduce DBS-induced speech disorders with the help of automated acoustic analysis in patients with STN-DBS-induced dysarthria.

In Part 1, the investigators' aim is to identify the most sensitive and specific speech variables for STN-DBS-related improvement of parkinsonian dysarthria and STN-DBS-induced speech-related side-effects, by application of an automated acoustic speech analysis technique. Patients with STN-DSB induced dysarthria will be examined in their medication ON state. Where possible the study will also be performed in the medication OFF state (after an overnight withdrawal of their PD medication). In both states, speech analysis will be performed in the stimulation OFF and ON states, as well as with increasing stimulation amplitudes.

In Part 2, the investigators' aim at investigating the anatomical and pathophysiological substrates of STN-DBS induced changes in speech production, by establishing stimulation maps. Stimulation maps highlight effective regions of stimulation and can help clinicians to navigate and program DBS steering the current towards the target region that improves speech (here a priori the sensorimotor STN for improving parkinsonian speech together with other parkinsonian signs), while avoiding current diffusion to regions identified as potentially worsening speech.

Part 3 is explorative. The investigators' hypothesize, that selected speech variables in automated speech analysis (as identified in part 1+2) are more sensitive to improvement of STN-DBS induced dysarthria, than ratings of three blinded speech-therapists. Again patients with STN-DBS induced dysarthria will be recruited to this study (willing participants of part 1+2 and patients who did not participate in part 1+2 will be included). The investigators will assess dysarthria by automated speech analysis, expert ratings and subjective ratings, before (at baseline visit) and at two time points (at V1 between 0-6 weeks after baseline and at V2 between 6-12 weeks after V1) after measures are taken to reduce stimulation induced dysarthria. Measures to reduce STN-DBS induced dysarthria will include all DBS settings that are routinely applied in daily clinical practice for dysarthria reduction. DBS-settings will be performed on both DBS-leads and patients will be in the medication ON state.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson-Syndrome according to the Movement Disorders Society Criteria
* Treatment with bilateral deep brain stimulation in the subthalamic nucleus (for parts 1, 2 and 3)
* Time since DBS-STN operation ≥ 3 month (for parts 1, 2 and 3)
* Able to give informed consent as documented by signature
* Fluent in Swiss-German or German
* STN-DBS-induced dysarthria. In an operational definition, all PD-patients who reported -worsening of speech time-locked to STN-DBS implantation or patients with dysarthria on chronic stimulation improving with reduction of stimulation amplitudes in the context of postoperative routine follow up will be defined as having STN-DBS-induced dysarthria

Exclusion Criteria:

* Dysarthria caused in addition by a condition other than PD or DBS (e.g. stroke, myasthenia)
* Clinical diagnosis of aphasia
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders and dementia. A Montreal Cognitive Assesment (MoCa) will be performed and patients with ≤ 20 of 30 points will be excluded
* Change of parkinsonian medication in the last four weeks prior to inclusion in part 1 and 3
* Change of STN-DBS parameters in the last four weeks prior to inclusion (for parts 1 and 3)
* Depression with acute suicidal ideation
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Part 1: Identification of the most sensitive and specific speech variables | At visit 1 (baseline visit)
  Identification of the most sensitive and specific speech variables of an automated acoustic analysis method, for STN-DBS-related improvement as well as worsening of speech in PD patients, under the two conditions (dopaminergic ON and OFF drug state).
  Speech variables will be extracted from the automated acoustic analysis.
Part 1: Identification of the most sensitive and specific speech variables | At visit 2 (≤4 weeks after visit 1)
  Identification of the most sensitive and specific speech variables of an automated acoustic analysis method, for STN-DBS-related improvement as well as worsening of speech in PD patients, under the two conditions (dopaminergic ON and OFF drug state).
  Speech variables will be extracted from the automated acoustic analysis.
Part 2, Speech analysis: Investigation of spatial overlap of volume of tissue activated (VTA) and the corticobulbar/corticospinal tract | 12 months
  Investigation of spatial overlap of tissue activated (VTA) and the corticobulbar/corticospinal tract, in relation to the dysarthria-worsening.
Part 2, Speech analysis: Investigation of spatial overlap of VTA and the dorsolateral (sensorimotor) STN | 12 months
  Investigation of spatial overlap of VTA and the dorsolateral (sensorimotor) STN in relation to improvement of PD-related dysarthria.
Part 3: Perceptual speech ratings | At baseline visit
  To test if the model 'perceptual speech ratings' explains subjective improvement of STN-DBS induced dysarthria.
  Perceptive rating will be performed by three experienced speech therapists, who will rate speech on a visual analogue scale (VAS).
Part 3: Perceptual speech ratings | At visit 1 (0-6 weeks after baseline)
  To test if the model 'perceptual speech ratings' explains subjective improvement of STN-DBS induced dysarthria.
  Perceptive rating will be performed by three experienced speech therapists, who will rate speech on a visual analogue scale (VAS).
Part 3: Perceptual speech ratings | At visit 2 (6-12 weeks after visit 1)
  To test if the model 'perceptual speech ratings' explains subjective improvement of STN-DBS induced dysarthria.
  Perceptive rating will be performed by three experienced speech therapists, who will rate speech on a visual analogue scale (VAS).
Part 3: Automated speech analysis | At baseline visit
  To test if the model 'automated speech analysis' explains subjective improvement of STN-DBS induced dysarthria.
  From the automated speech analysis, only the speech parameters explaining most of the variance in the model from part 2 will be included in the analysis.
Part 3: Automated speech analysis | At visit 1 (0-6 weeks after baseline)
  To test if the model 'automated speech analysis' explains subjective improvement of STN-DBS induced dysarthria.
  From the automated speech analysis, only the speech parameters explaining most of the variance in the model from part 2 will be included in the analysis.
Part 3: Automated speech analysis | At visit 2 (6-12 weeks after visit 1)
  To test if the model 'automated speech analysis' explains subjective improvement of STN-DBS induced dysarthria.
  From the automated speech analysis, only the speech parameters explaining most of the variance in the model from part 2 will be included in the analysis.

SECONDARY OUTCOMES:
Part 1: Subjective rating of the quality of speech | At visit 1 (baseline visit) and visit 2 (≤4 weeks)
  Subjective rating of the quality of speech on a numeric rating scale by the patient, ranging from 0 = no impairment to 10 = maximum conceivable impairment of speech. Assessment will be performed under the two conditions (dopaminergic ON and OFF drug state).
Part 1: Assessment parkinsonism contralateral to the tested DBS lead | At visit 1 (baseline visit) and visit 2 (≤4 weeks)
  Assessment parkinsonism contralateral to the tested DBS lead using items 3.4 (finger tapping), 3.5 (hand movements), 3.7 (toe tapping) and 3.8 (leg agility) of the Movement Disorders Society-Unified Parkinson's Disease Rating Scale part III (MDS-UPDRS part III) for the limbs contralateral to the tested DBS electrode. Assessment will be performed under the two conditions (dopaminergic ON and OFF drug state).
Part 1: Clinical assessment of possible side effects | At visit 1 (baseline visit) and visit 2 (≤4 weeks)
  Noting possible side effects that may occur during the experiment, such as fascial spasm or contraction of the hand muscles. Assessment will be performed under the two conditions (dopaminergic ON and OFF drug state).
Part 3: Subjective rating of the quality of speech | At baseline visit, visit 1 (0-6 weeks after baseline) and visit 2 (6-12 weeks after visit 1)
  Subjective rating of the quality of speech on a numeric rating scale by the patient, ranging from 0 = no impairment to 10 = maximum conceivable impairment of speech.
Part 3: Assessment of motoric symptoms | At baseline visit, visit 1 (0-6 weeks after baseline) and visit 2 (6-12 weeks after visit 1)
  Assessment of Parkinsonism using the full Movement Disorders Society-Unified Parkinson's Disease Rating Scale part III (MDS-UPDRS part III).
Part 3: Clinical assessment of possible side effects | At baseline visit, visit 1 (0-6 weeks after baseline) and visit 2 (6-12 weeks after visit 1)
  Noting possible side effects that may occur during the experiment, such as fascial spasm or contraction of the hand muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Krack, Prof., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (2):
- Czech Technical University Prague, Prague, Czechia
- University Hospital Inselspital, Berne, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No